CLINICAL TRIAL: NCT04932759
Title: Investigation Of The Effect Of Music Listened By Patients With Moderate Dental Anxiety During The Restoration Of Posterior Occlusal Dental Caries
Brief Title: The Effect Of Music Listened By Patients With Moderate Dental Anxiety During The Restoration Of Occlusal Caries
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karadeniz Technical University (Other)
Responsible Party: Principal Investigator, Kıvanc Dulger, Assistant Professor, Karadeniz Technical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2020-41
Record Dates: First submitted 2021-06-05; First posted 2021-06-21 (Actual); Last update posted 2023-10-05 (Actual); Status verified 2023-10

CONDITIONS: Dental Anxiety; Music; Physical Stress
Keywords: dental anxiety; music

STUDY DESIGN:
Intervention Model Description: Control and study group
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group (No Intervention): In the control group there will be no music listening
- experimental group (Experimental): In this group patients will listen to music while their dental treatments are being made.
  Interventions: Behavioral: music listening

INTERVENTIONS:
Behavioral: music listening — music listening during dental treatment
  Arms: experimental group

SUMMARY:
It is aimed to evaluate the effect of music listened by patients with moderate dental anxiety during the restoration of posterior occlusal dental caries on vital signs of the participants.

DETAILED DESCRIPTION:
The study will be applied on 70 patients; 35 patients will be in the control group (the group not listening to music during treatment), 35 patients will be in the experimental group (the group listening to music during treatment).

Modified Dental Anxiety Scale consisting of 5 questions will be applied to the participants who come to the clinic and have occlusal dental caries in the posterior region. The participants whose scores are between 10-18 according to this scale will be included in the study. One occlusal tooth decay will be treated. Before starting treatment, saliva cortisol levels, heart rate, body temperature, systolic and diastolic blood pressure and oxygen saturation measurements will be made. The participants will be asked to spit in sterile plastic containers for saliva cortisol measurement. During dental treatment, the participants will listen to music in experimental group. In control group the participant will not listen to music. Heart rate, body temperature, systolic and diastolic blood pressure and oxygen saturation measurements will be repeated in the middle of the treatment (without going through the restoration phase when the cavity is opened). Saliva cortisol levels, heart rate, body temperature, systolic and diastolic blood pressure and oxygen saturation measurements will be repeated when the treatment is completed. The questionnaire containing the modified dental anxiety scale will be re-administered to the participants.

ELIGIBILITY:
Inclusion Criteria:

Must be healthy volunteers, Clinical diagnosis of at least one occlusal dental caries, Must have moderate dental anxiety

-

Exclusion Criteria:Unhealthy volunteers, Teeth with dental cavities in the adjacent teeth where the rubber dam would not be placed, and dental caries closer than 1 mm to the pulp tissue were not included in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2021-01-10 (Actual); Primary Completion 2021-12-10 (Actual); Study Completion 2022-01-10 (Actual)

PRIMARY OUTCOMES:
Salivary cortisol level | Before-after
  Change of salivay cortisol level (before-after)
Vital anxiety signs | Before-after
  Change of heart rate, body temperature, systolic and diastolic blood pressure and oxygen saturation measurements

SECONDARY OUTCOMES:
Modified dental anxiety questionnaire | Before-after
  Modified dental anxiety questionnaire will be applied to participants after finishing dental treatment

CONTACTS AND LOCATIONS:
Overall Officials: KIVANÇ DÜLGER, Study Director — Asst Prof
Locations (1):
- Karadeniz Technical University Faculty of Dentistry, Trabzon, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
After the completing of the study, the data will be written as a research article.

REFERENCES:
- [Background] Aravena PC, Almonacid C, Mancilla MI. Effect of music at 432 Hz and 440 Hz on dental anxiety and salivary cortisol levels in patients undergoing tooth extraction: a randomized clinical trial. J Appl Oral Sci. 2020;28:e20190601. doi: 10.1590/1678-7757-2019-0601. Epub 2020 May 11. PMID 32401941
- [Background] Mejia-Rubalcava C, Alanis-Tavira J, Mendieta-Zeron H, Sanchez-Perez L. Changes induced by music therapy to physiologic parameters in patients with dental anxiety. Complement Ther Clin Pract. 2015 Nov;21(4):282-6. doi: 10.1016/j.ctcp.2015.10.005. Epub 2015 Oct 27. PMID 26573456
- [Background] Bradt J, Teague A. Music interventions for dental anxiety. Oral Dis. 2018 Apr;24(3):300-306. doi: 10.1111/odi.12615. Epub 2017 Jan 5. PMID 27886431